CLINICAL TRIAL: NCT02002585
Title: Renal Protection Using Sympathetic Denervation in Patients With Chronic Kidney Disease (Kidney Protection Study - KPS Study)
Brief Title: Renal Protection Using Sympathetic Denervation in Patients With Chronic Kidney Disease
Acronym: KPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other); Na Homolce Hospital (Other); Mount Sinai Hospital, New York (Other)
Responsible Party: Principal Investigator, Ass. prof. Jean-Claude M. Lubanda, MD, Ph.D, Associate professor, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPS1
Record Dates: First submitted 2013-11-25; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Arterial Hypertension; Chronic Renal Insufficiency
Keywords: Renal protection; Renal sympathetic denervation
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RDN and optimal medical therapy (Experimental): Renal denervation will be performed using the available denervation device with a european approval according to current guidelines. The same device will be used for all patients in this arm to avoid efficacy bias.
  Interventions: Procedure: Renal denervation
- optimal medical therapy alone (No Intervention): Group of patients who will be treated only with optimal medical therapy and will not be denervated. Subsequently, the patients will be followed in our cardiology and nephrology department according to the study flowchart for 3 years according to the standard of care in our institution for patients with chronic renal insufficiency.

INTERVENTIONS:
Procedure: Renal denervation — Catheter based renal sympathetic denervation is a endovascular method used for the treatment of resistent hypertension.
  Other Names: RDN - Renal sympathetic denervation
  Arms: RDN and optimal medical therapy

SUMMARY:
Kidney protection study (KPS 1) is a prospective randomized clinical study comparing the use of renal denervation (RDN) and optimal medical therapy in subjects with chronic kidney disease stage 3-4 and resistant arterial hypertension to optimal medical therapy alone. Renal denervation is a modern endovascular method used to treat resistant hypertension. The method is being extended to other groups of patients, where the sympathetic tone is increased beyond resistant hypertension. Because of the character of the disease, we hypothesize that renal denervation can reduce or prevent progressive deterioration of kidney functions in this patient population. The aim of this clinical study is to show that renal denervation has protective effects on the progression of chronic renal insufficiency.

DETAILED DESCRIPTION:
Background:

patients with chronic renal insufficiency are an ideal group for renal denervation (RDN), because of the increase in sympathetic tone. This increase leads to sodium retention, reduction of perfusion of the kidney and to excessive activation of renin angiotensin aldosterone system. The activation of the sympathetic system significantly contributes to the progression of chronic renal insufficiency. The consequences the hyperactivity of the sympathetic system are affected by selective renal sympathectomy. RDN demonstrably reduces retention of sodium, reduces the production of renin and significantly reduces renal vascular resistance. Furthermore, RDN reduces microalbuminuria and renal podocyte damage in experimental model. RDN also improves renal function in the model of acute Glomerulonephritis. In patients with resistant hypertension and preserved renal function, it was also shown that renal denervation improves renal resistant index and significantly decreases microalbuminuria. The procedure was found to be safe in all studies with renal denervation and was not associated with deterioration of renal function. Several experimental data exist on the effectiveness of RDN in chronic renal insufficiency. In a model of acute renal failure in mouse (endotoxemia model), it was shown that RDN has protective effect on renal function. The decline in the glomerular filtration during endotoxemia was significantly lower in the group treated with RDN compared to the control group. In addition, the renal flow during acute renal failure after RDN was improved. In the model of heart failure in mice, it has been shown that RDN in combination with olmesartan reduces albuminuria and the damage of podocytes and also reduces the levels of renal norepinephrine, angiotensinogen, angiotensin II, and the level of oxidative stress.

Very few data on the effect of RDN on renal function in human were also published. Renal damage in hypertensives subject was not found after RDN with the Symplicity system more than 3 years post procedure. Mahfoud and coworkers showed that subject treated with RDN had lower blood pressure and renal resistive index and at the same time stabilize their renal function. The number of patients with microalbuminuria or macroalbuminuria decreased significantly one year after RDN.

RDN has also positive effect on albuminuria and proteinuria in patients with preserved renal function. The first studies performed in patients with chronic kidney disease (CKD stage 3-4) and resistant hypertension was done by Hering et coworkers. In this study, 15 patients with an average eGFR of 31ml/min/1, 73m2 underwent RDN. The authors were able to show that RDN effectively lowers blood pressure and was not associated further deterioration of renal function. RDN had other positive effects on hemoglobin concentration , proteinuria and on BNP levels. Moreover, the augmentation index of peripheral arteries was also improved by RDN. This work showed multiple effects of RDN beyond the reduction of blood pressure. We, therefore think that patient with chronic kidney disease are good candidates for RDN. However, the mentioned study has a relatively short term follow up (6 months to one year) and does not have a comparative arm.

Aim of study :

our proposed trial aimed to show that RDN not only contribute to improve the control of blood pressure in patients with resistant hypertension but also has protective effects on kidney function in subjects with chronic kidney disease. Our trial will have a comparative arm and will last 3 years.

Planned intervention:

The two strategies that are going to be compared are optimal medical therapy against optimal medical therapy with renal denervation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18-80 years
* Chronic renal insufficiency in CKD 3-4 from nephrologist (eGFR (MDRD) ≤ 45 ml/min/1.73 m2)
* Arterial hypertension treated with:

systolic BP ≥ 140 mmHg + at least 3 antihypertensive drugs Including a diuretic systolic BP ≥ 135 mmHg + 3 antihypertensives Including a diuretics + diabetes mellitus type 2.

systolic BP ≥ 130 mmHg on 24 hr ABPM + 3 antihypertensive drugs Including a diuretics

• Renal artery diameter ≥ 4 mm according to the renal angiography (documented on quantitative renal angiography), renal artery length at least 20mm

Exclusion Criteria:

* Secondary hypertension
* White coat hypertension
* abnormalities in renal angiogram disqualifying for RDN
* Life expectancy < 1 year
* Type 1. Diabetes mellitus
* Significant stenotic valvular heart disease
* Acute coronary syndrome of unstable angina in the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The changes of eGFR by MDRD | 6 months
  The changes of the value of eGFR measured using the MDRD equation in both groups measure at baseline and after 6 months
Changes in proteinuria (Microalbuminuria) in 6 months | 6 months
  the change in the value of proteinuria expressed in g/24hrs or microalbuminuria expressed in ug/24hrs measured at baseline compared to value at 6 month in both study groups
Changes in the value of Cystatin C | 6 months
  Changes in the value of Cystatin C measure at baseline and after 6 months in both groups
Time to the development of end-stage renal disease (ESRD)/Hemodialysis | 3 years
  The time to the development of end-stage renal disease (ESRD)/Hemodialysis in both groups
combined renal endpoint | 6 months
  the combination of all primary outcomes measured compared to baseline in both groups

SECONDARY OUTCOMES:
Total mortality | 3 years
  the total mortality in both groups at 6 months, 2 years and 3 years
The total cardiovascular mortality | 3 years
  the total cardiovascular mortality in 6 months, 2 years and 3 years in both groups
total renal mortality | 3 years
  the total renal mortality in both arms at 6 months, 2 years and 3 years
changes in blood pressure | 3 years
  the changes of systolic and diastolic blood pressure at 6 months, 1, 2 and 3 years measured as office blood pressure, home blood pressure monitoring and ambulatory blood pressure monitoring (ABPM) from baseline in both arms
•Changes in concentration of Blood urea Nitrogen (BUN) , creatinine in 6 months, 3 years | 3 years
  the changes in concentration of blood urea Nitrogen (BUN) and creatinine in 6 months, 1, 2 and 3 years in both arms
albumin-creatine ratio | 3 years
  Albumin-Creatinine-Ratio (mg/mmol) in 6 months, 1, 2 and 3 years in both arms
changes in cardiac structure and function | 3 years
  the changes in cardiac structure and function assessed by echocardiography (left ventricular mass, left ventricular ejection fraction, left ventricular diastolic function) at 6 months, 1, 2 and 3 years in both arms.
the changes in renal resistive index | 3 years
  •the changes in renal resistive index (RRI) measured using renal duplex ultrasound at 6 months, 1, 2 and 3 years in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Jean Claude Lubanda, Ass.Prof. MD, Principal Investigator — Charles University, Czech Republic
Locations (1):
- Charles University in Prague, Prague, Czechia